CLINICAL TRIAL: NCT04674241
Title: Effect of Dexmedetomidine on Postoperative Delirium in Patients Undergoing Brain Tumor Resections: a Randomized Controlled Study
Brief Title: Dexmedetomidine Alleviates Postoperative Delirium After Brain Tumor Resections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Deputy chief of Department of Anethesiology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ChiECRCT20200436
Record Dates: First submitted 2020-12-13; First posted 2020-12-19 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Dexmedetomidine; Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX group (Active Comparator): The DEX group will receives dexmedetomidine intraoperative.
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): The placebo group will receives 0.9% saline intraoperative.
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Dexmedetomidine — Ten minutes after anesthesia induction and endotracheal intubation, patients assigned to dexmedetomidine group were given a loading dose of dexmedetomidine 0.6 μg/kg over 10 minutes, followed by continuous infusion at a rate of 0.4 μg/kg/h until the start of dural closure.
  Arms: DEX group
Drug: 0.9% saline — 0.9% saline is administered with the same volume at the same speed as the other group.
  Arms: Placebo group

SUMMARY:
Postoperative delirium (POD) is a common complication, and the incidence rate is about 25% in non cardiac surgery. Previous studies have reported that the total incidence of neurological pod ranged from 10% to 22%. Dexmedetomidine (DEX) is an a-2 adrenergic agonist for sedation. This kind of drug has little effect on respiratory function, is easy to wake up and has analgesic effect. It is a commonly used perioperative adjuvant drug. However, for neurosurgical patients with brain tumors, the role of DEX in POD is not clear. The purpose of this study was to investigate the effect of DEX on POD in neurosurgical brain tumor surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing selective frontotemporal tumor resection.
* Age ≥18 years.
* Obtain written informed consent.

Exclusion Criteria:

* Refusal to provide written informed consent.
* Preoperative severe cognitive impairment (mini-mental state examination, MMSE ≤ 20).
* Allergic to the study drug.
* History of psychotropic drugs within past 30 days.
* Pregnant or lactating women.
* History of traumatic brain injury or neurosurgery.
* Severe bradycardia (heart rate less than 40 beats per minute), sick sinus syndrome or second-to-third degree atrioventricular block.
* Severe hepatic or renal dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative delirium | postoperative 5 day
  Postoperative delirium is assessed by the combination of the Richmond Anxiety Scale (RASS) and the Confusion assessment method for intensive care unit (CAM-ICU) or the 3-minute diagnostic interview for CAM (3D-CAM) as applicable.
  Delirium consists of four main characteristics: acute onset of a change in mental status or a fluctuating level of consciousness, inattention, disorganized thinking and an altered level of consciousness. The patient was diagnosed as delirious if both the first and second features were present, and either the third or fourth was present.
  In the ICU, the delirium assessment was performed in two steps. The arousal level was first assessed by RASS. If the patient was not responsive to verbal stimuli (i.e. RASS score ≤-4), the remaining delirium assessment was aborted, and the patient was recorded as comatose. When the RASS score was greater than or equal to 3, delirium was evaluated using the CAM-ICU. Patients in general ward were evaluated by 3D-CAM.

SECONDARY OUTCOMES:
Pain score | within 5 days after surgery
  Numerical Rating Scales, ranging from 0 to 10 points, with 10 representing the worst imaginable pain.
Sleep quality | within 3 days after surgery
  Quality of sleep was assessed by the Richards Campbell sleep questionnaire (RCSQ) and with a 0-100-mm visual analog scale, with higher scores indicating better sleep quality.
Quality of recovery from surgery | 1 day after surgery
  Postoperative quality of recovery was assessed through the Quality of Recovery 15 item
Intraoperative cardiovascular event. | From the study drug infusion to the end of surgery.
  Including: hypotension was defined as systolic blood pressure <95 mm Hg or less than 30% below baseline; hypertension was defined as systolic blood pressure > 180 mm Hg or more than 30% above baseline; bradycardia was defined by heart rate <40 bpm, and tachycardia was defined by heart rate >100 bpm.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Ming Peng, MD,Ph.D, Principal Investigator — Beijing Tian Tan Hospital
Locations (2):
- China (2):
  - Beijing TianTan Hospital,Capital Medical University, Beijing, Beijing,China
  - PLA General Hospital, Beijing

REFERENCES:
- [Derived] Wu Y, Ren Y, Li S, Zeng M, Wang J, Li M, Peng Y. Association between intraoperative hypotension during brain tumor resection and postoperative delirium: A secondary analysis of a randomized controlled trial. PLoS One. 2025 Oct 29;20(10):e0334094. doi: 10.1371/journal.pone.0334094. eCollection 2025. PMID 41160633
- [Derived] Zeng M, Xu X, Li R, Zhang X, Ma T, Cui Q, Wang J, Li S, Peng Y. Dexmedetomidine Prevents Chronic Incisional Pain After Brain Tumor Resection: A Secondary Analysis of the Randomized Control Trial. Anesth Analg. 2024 Apr 1;138(4):839-847. doi: 10.1213/ANE.0000000000006563. Epub 2023 Jun 12. PMID 37307232
- [Derived] Li S, Li R, Li M, Cui Q, Zhang X, Ma T, Wang D, Zeng M, Li H, Bao Z, Peng Y, Sessler DI. Dexmedetomidine administration during brain tumour resection for prevention of postoperative delirium: a randomised trial. Br J Anaesth. 2023 Feb;130(2):e307-e316. doi: 10.1016/j.bja.2022.10.041. Epub 2022 Dec 13. PMID 36517290
- [Derived] Wang D, Li R, Li S, Wang J, Zeng M, Dong J, Liu X, Lin N, Peng Y. Effect of dexmedetomidine on postoperative delirium in patients undergoing brain tumour resections: study protocol of a randomised controlled trial. BMJ Open. 2021 Nov 10;11(11):e051584. doi: 10.1136/bmjopen-2021-051584. PMID 34758995